CLINICAL TRIAL: NCT07381400
Title: A Multicenter, Randomized Controlled Clinical Study of Neoadjuvant mFOLFOX6 Chemotherapy Combined With Anti-PD-1 Therapy in MSS/pMMR Locally Advanced Rectal Cancer (FIRM02 Study)
Brief Title: Neoadjuvant mFOLFOX6 Chemotherapy Combined With Anti-PD-1 Therapy in MSS/pMMR Locally Advanced Rectal Cancer (FIRM02 Study)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Tingyu Wu, Dr., Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2025-300-2
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; PD1 inhibitor; pMMR; microsatellite stable; neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOX6+Serplulimab (Experimental): Preoperative treatment with mFOLFOX6 chemotherapy combined with Serplulimab (3mg/kg) every 2 weeks, for a total of 6 cycles before surgery.
  Interventions: Drug: mFOLFOX6; Drug: Serplulimab
- mFOLFOX6 (Active Comparator): Preoperative treatment with mFOLFOX6 chemotherapy every 2 weeks, for a total of 6 cycles before surgery.
  Interventions: Drug: mFOLFOX6

INTERVENTIONS:
Drug: mFOLFOX6 — Oxaliplatin 85 mg/m², intravenous infusion on Day 1; Fluorouracil 400 mg/m², intravenous infusion on Day 1; Fluorouracil 2400 mg/m², continuous infusion via chemotherapy pump for 46-48 hours; Leucovorin calcium 400 mg/m², intravenous infusion on Day 1 (or Levoleucovorin 200 mg/m², intravenous infusion).
Drug: Serplulimab — 3 mg/kg, intravenous infusion, Day 1.
  Arms: mFOLFOX6+Serplulimab

SUMMARY:
This multicenter, randomized controlled clinical trial (FIRM02 Study) aims to evaluate the effectiveness and safety of neoadjuvant mFOLFOX6 chemotherapy combined with PD-1 inhibitor (Serplulimab) in patients with MSS/pMMR locally advanced rectal cancer (LARC). A total of 128 patients with non-metastatic, untreated, locally advanced rectal cancer will be randomly assigned in a 1:1 ratio to either the experimental group (64 patients) or the control group (64 patients). The experimental group will receive 6 cycles of mFOLFOX6 chemotherapy combined with 3 mg/kg of Serplulimab every 2 weeks prior to surgery. The control group will receive 6 cycles of mFOLFOX6 chemotherapy alone. The primary endpoint is the pathological complete response (pCR), and secondary endpoints include major pathological response (MPR), tumor regression grade (TRG), overall response rate (ORR), and survival outcomes (DFS, RFS, and OS). Safety will be assessed based on adverse events and post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Rectal cancer patients with MRI showing the lower edge of the tumor within 15 cm of the anal verge, cT3-4 N any or cT any N1/2;
2. Pathologically confirmed adenocarcinoma, with pMMR (MLH1, MSH2, MSH6, and PMS2) positivity for all four proteins, or gene testing indicating microsatellite stability;
3. No complete bowel obstruction, or proximal colostomy relieving bowel obstruction;
4. Aged 18 to 75 years, regardless of gender;
5. ECOG performance status: 0-1;
6. Expected survival time ≥2 years;
7. No previous chemotherapy, radiotherapy, targeted therapy, or immunotherapy;
8. Laboratory test results meeting the following criteria during screening:Hematology: Neutrophil count ≥1.5×10⁹/L, platelet count ≥75×10⁹/L, hemoglobin ≥80 g/L; Liver function: AST and ALT ≤2.5× upper limit of normal (ULN); total bilirubin ≤1.5×ULN; Kidney function: Serum creatinine ≤1.5×ULN; Coagulation function: APTT ≤1.5×ULN, INR ≤1.5, PT ≤1.5×ULN; Urine protein: Urine protein ≤1+ (if ≥2+, 24-hour urine protein test required, and if result <1g, inclusion is allowed); Cardiac left ventricular ejection fraction ≥50%;
9. Female participants must not be breastfeeding, and pregnancy test results must be negative;
10. Voluntary signing of the informed consent form, with the ability to understand and comply with the study requirements.

Exclusion Criteria:

1. Local invasion of surrounding organs by rectal tumor: Imaging tests suggest the tumor directly invades adjacent organs or structures, i.e., tumors with clinical stage cT4 below the peritoneal reflection or cT4b above the peritoneal reflection;
2. Patients with distant metastasis;
3. Previous treatment with any chemotherapy, radiotherapy, targeted therapy, or immunotherapy;
4. Active autoimmune diseases requiring systemic treatment (e.g., corticosteroids or immunosuppressants) within the past 2 years prior to enrollment;
5. History of HIV infection, or active chronic hepatitis B or C (high viral DNA load);
6. Currently receiving tuberculosis treatment or having received tuberculosis treatment in the past year prior to screening for active tuberculosis;
7. Known or suspected allergy to the study drugs or any drug related to the study;
8. Severe cardiovascular or cerebrovascular diseases;
9. Severe active infection or uncontrollable infection requiring systemic treatment, or unexplained fever >38.5°C within 14 days before the first dose;
10. Systemic corticosteroid treatment or other immunosuppressants within 14 days before the first dose, or immunostimulants within 4 weeks prior to the first dose;
11. Clear history of neurological or psychiatric disorders, including epilepsy or dementia;
12. Subjects who, for any other reason, may not be able to complete the study, or the investigator deems them unsuitable for inclusion;
13. Refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response Rate (pCR) | Day 7 after surgery

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | Day 7 after surgery
Tumor regression grade | Day 7 after surgery
Objective Response Rate | Pre-neoadjuvant therapy, Post-neoadjuvant therapy.
Neoadjuvant rectal score | Day 7 after surgery
  The Neoadjuvant Rectal Score (NAR) ranges from 0 to 100, with lower scores indicating better neoadjuvant efficacy.
R0 resection rate | Day 7 after surgery
Sphincter preservation rate | Surgical date
Overall Survival | Five years after surgery
Recurrence-Free Survival | Five years after surgery
Disease-Free Survival | Five years after surgery
Treatment-Related Adverse Events | Adverse events are evaluated the day before each chemotherapy cycle, up to 90 days after the last neoadjuvant treatment.
Surgical-related complications | Within 1 month post-surgery

IPD SHARING:
Plan to Share IPD: Yes
In this study personal information and data such as patient history, physical examination results, surgical records, and study questionnaire data will be collected. These data will be used to evaluate the efficacy and safety of the therapeutic regimen and for academic publication. The researcher will treat the personal data of patients confidentially and anonymize the data and information in any public release of the results of the study.
Supporting Information: Study Protocol, SAP